CLINICAL TRIAL: NCT04163198
Title: Investigating Methods to Improve Secretion Clearance Using Mechanical Insufflation:Exsufflation in Patients With Neuromuscular Disease.
Brief Title: Optimisation of Mechanical Insufflation:Exsufflation
Acronym: MIE2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Insufflation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insufflation optimisation (Experimental): Patient will receive different inspiratory time and expiratory time, and inspiratory flow at a fixed insufflation pressure. To determine how best to recruit lung.
  Interventions: Device: Insufflation
- Exsufflation optimisation (Experimental): Patient will receive different expiratory pressures at a fixed inspiratory pressure (optimal determine in Arm 1). To determine minimum flow bias needed to generate cPEF
  Interventions: Device: Exsufflation

INTERVENTIONS:
Device: Insufflation — Patients will receive different inspiratory (Ti) and expiratory (Te) times and inspiratory flows, at a fixed insufflation and exsufflation pressure. Optimum insufflation pressure will be determined by measuring maximal inspiratory capacity.
  Arms: Insufflation optimisation
Device: Exsufflation — Patients will receive different exsufflation pressures at fixed insufflation pressure.
  Arms: Exsufflation optimisation

SUMMARY:
Patients with neuromuscular diseases (NMD) can suffer from a range of respiratory problems due to respiratory muscle weakness. Cough muscle weakness means secretion clearance from the airways can be problematic, a source of infection, and importantly a cause of death, in this patient group. Therefore, these patients are often supported with devices to aid clearance, such as mechanical insufflation-exsufflation (MIE). Although evidence supports the use of these devices, the optimal technique or settings on the device are not clear. Increasingly, higher pressures are used during MIE and recent work has demonstrated that there may be a physiological benefit to this. However, higher pressures increase the risk of causing lung collapse and may cause detriment to blood flow back to the heart, which is important as NMD patients frequently have concurrent heart muscle weakness. Further, recent work has demonstrated that higher pressures can cause closure of the throat, which is counter-productive in secretion clearance.

The overall aim of this study is to investigate methods to manipulate MIE to improve secretion clearance in patients with NMD. The questions it seeks to answer are:

(i) how can we maximally improve lung recruitment during inspiration, whilst maintaining patient comfort and lower pressures (ii) what is the smallest pressure difference required in expiration to achieve an improvement in cough (iii) do these proposed changes to MIE also cause throat closure (iv) what factors do patients believe contribute to their adherence to MIE therapy?

Patients with slowly progressive or stable neuromuscular diseases will be included in the study. Participation will involve two visits to the Lane Fox Respiratory Unit, each lasting approximately four hours. Patients will be recruited from specialist neuromuscular respiratory clinics by their clinical teams.

ELIGIBILITY:
Inclusion Criteria:

* Stable or slowly progressive neuromuscular disease
* Respiratory muscle weakness (FVC <60%, snip <60%, sleep disordered breathing)
* Clinical evidence of respiratory secretions or cough peak expiratory flow <270 and history of lower respiratory tract infection
* Documented clinical stability by supervising clinician

Exclusion Criteria:

* Rapidly progressive neuromuscular disease (such as motor neuron disease)
* Decompensated respiratory failure (pH < 7.35)
* Pregnancy
* Aged <18
* Change in ventilator settings in preceding 4 weeks
* Significant physical or psychiatric co-morbidity that would prevent compliance with trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Cough peak expiratory flow (cPEF) | 2 days
  Change in cPEF with different modalities of MI-E

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Murphy, PhD, Study Chair — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys & St. Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No